CLINICAL TRIAL: NCT00546585
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase I/II, Dose-Ranging Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H7N7 Vaccine in Healthy Adults
Brief Title: Safety, Reactogenicity, and Immunogenicity of Inactivated Influenza A/H7/N7 Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-0023
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2010-01

CONDITIONS: Influenza
Keywords: influenza, inactivated influenza A/H7N7 vaccine, parent protocol
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- 90 mcg of Influenza A/H7N7 (Experimental): 25 subjects to receive 90 mcg of Influenza A/H7N7.
  Interventions: Biological: Influenza A/H7N7 Vaccine
- 15 mcg of Influenza A/H7N7 (Experimental): 25 subjects to receive 15 mcg of Influenza A/H7N7.
  Interventions: Biological: Influenza A/H7N7 Vaccine
- 7.5 mcg of Influenza A/H7N7 (Experimental): 25 subjects to receive 7.5 mcg of Influenza A/H7N7.
  Interventions: Biological: Influenza A/H7N7 Vaccine
- 45 mcg of Influenza A/H7N7 (Experimental): 25 subjects to receive 45 mcg of Influenza A/H7N7.
  Interventions: Biological: Influenza A/H7N7 Vaccine
- Saline placebo (Placebo Comparator): 25 subjects to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Influenza A/H7N7 Vaccine — Monovalent subvirion H7N7 vaccine, 4 dose levels of vaccine, each subject will receive 2 doses (7.5, 15, 45, or 90 micrograms); the same dose will be given at Day 0 and Day 28.
  Arms: 15 mcg of Influenza A/H7N7; 45 mcg of Influenza A/H7N7; 7.5 mcg of Influenza A/H7N7; 90 mcg of Influenza A/H7N7
Drug: Placebo — Sterile normal saline for injection (0.9%); 0.5 ml volume sodium chloride injection. Subjects will receive 2 doses on Day 0 and Day 28.
  Arms: Saline placebo

SUMMARY:
The purpose of this study is to evaluate the safety, any adverse events or side effects, and the body's immune response to an experimental flu vaccine [Inactivated Influenza A/H7N7 Vaccine] being given in increasing doses. Researchers will try to find the smallest dose of flu vaccine needed to cause antibody responses against the flu virus in both single and repeat doses. The study will enroll 125 healthy adults ranging in age from 18 to 40 years old. Subjects will be given 2 doses of the vaccine 28 days apart. Study procedures will include obtaining a medical history, physical exam, blood sample collections, and use of patient memory aids. The volunteers will be in the study for about 7 months.

DETAILED DESCRIPTION:
This randomized, double-blinded, placebo-controlled, dose-ranging, Phase I/II, influenza study will compare the safety, reactogenicity, and immunogenicity of increasing doses of monovalent subvirion influenza A/H7N7 virus vaccine administered by intramuscular (IM) injection to healthy adults. A total of 125 healthy adults ranging from 18 to 40 years old will be enrolled at one site for this study. The subjects will be randomized to receive saline placebo or 7.5, 15, 45, or 90 mcg of the influenza A/H7N7 vaccine by intramuscular (IM) injection in an approximate 1:1:1:1:1 ratio (N=25/vaccine dose group and 25 in the placebo group). Subjects will receive 2 doses separated by approximately 28 days. Subjects will be observed in the clinic for a minimum of 30 minutes after inoculation. All subjects will maintain a memory aid to record oral temperature and systemic and local adverse events (AEs) for 7 days after each immunization. Subjects will be contacted by telephone 1-3 days after vaccination to assess for the occurrence of AEs, and they will return to the clinic between Day 8 and 12 for AE and concomitant medication assessment, a targeted physical examination (if indicated), and review of the memory aid. Serum for immunogenicity evaluations will be obtained for subjects prior to the first vaccination, at Day 28 prior to the second vaccination, and on Days 56 and 208. A Safety Monitoring Committee (SMC) will review available 7 day safety data at approximately Day 20 following the first subject vaccination before administering the second dose of vaccine to any subjects. The primary objectives of the study will be: to determine the dose-related safety of subvirion inactivated H7N7 vaccine in healthy adults; to determine the dose-related immunogenicity of subvirion inactivated H7N7 vaccine in healthy adults approximately 1 month following receipt of 2 doses of vaccine; and to provide information for the selection of the best dose levels for further studies. The secondary objective will be to evaluate the dose-related immunogenicity and the percent of subjects responding approximately 1 and 7 months after the first vaccination. The primary endpoints are: adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessment); the proportion of subjects in each dose group achieving a serum neutralizing antibody titer of greater than or equal to 40 against the influenza A/H7N7 virus 28 days after receipt of the second dose of vaccine (approximately Day 56); geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 1 month after receipt of each dose, and 7 months after receipt of the first dose of vaccine; and GMT and frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) antibody titers in each group 1 month after receipt of each dose, and 7 months after receipt of the first dose of vaccine. Participants will be involved in study related procedures for approximately 7 months. This study is linked to DMID protocol 07-0060.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 40 years, inclusive.
* Women of childbearing potential (not surgically sterile or postmenopausal for greater than or equal to 1 year) who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier method, abstinence, intrauterine devices, and licensed hormonal methods) for the entire study period.
* Is in good health, as determined by vital signs (heart rate < 100 beats per minute, blood pressure: systolic less than or equal to 140 mm Hg and greater than or equal to 90 mm Hg, diastolic less than or equal to 90 mm Hg; oral temperature < 100 degrees Fahrenheit), medical history to ensure stable* medical condition and a targeted physical examination based on medical history. (*A stable medical condition is defined as no recent change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company, etc, or is done for financial reasons, as long as in the same class of medication, will not be considered a violation of the inclusion criterion. Any change to prescription medication due to improvement of a disease outcome will not be considered a violation of the inclusion criterion.)
* Able to understand and comply with planned study procedures.
* Provide informed consent prior to initiation of any study procedures and are available for all study visits.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol, aluminum hydroxide, and chicken protein).
* Have a positive urine or serum pregnancy test prior to vaccination (if female of childbearing potential) or women who are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed.)
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Have received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to vaccination in this study.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. (This includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* Have a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 1 week of vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study, or expect to receive an experimental agent during the 7-month study period.
* Plan to enroll in another clinical trial at any time during the study period.
* Have any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Have a diagnosis of schizophrenia, Bi-polar disease or other major psychiatric diagnosis.
* Have been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Are receiving psychiatric drugs*. Subjects who are receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.

  * aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate
* Have a known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Plan to travel outside of the USA in the time between the first vaccination and 56 days following the first vaccination.
* Have a history of Guillain-Barre syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessment). | Duration of study.
Proportion of subjects in each dose group achieving a serum neutralizing antibody titer of greater than or equal to 40 against the influenza A/H7N7 virus. | 28 days after receipt of the second dose of vaccine (approximately Day 56).
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group and serum hemagglutination inhibition (HAI) antibody titers in each group. | 1 month after receipt of each dose, and 7 months after receipt of the first dose of vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine - Department of Molecular Virology and Microbiology, Houston, Texas, United States

REFERENCES:
- [Result] Couch RB, Patel SM, Wade-Bowers CL, Nino D. A randomized clinical trial of an inactivated avian influenza A (H7N7) vaccine. PLoS One. 2012;7(12):e49704. doi: 10.1371/journal.pone.0049704. Epub 2012 Dec 11. PMID 23239968